CLINICAL TRIAL: NCT06792591
Title: Diagnostic Performance of Positron Emission Mammography in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zainab Fathy Mohammed, AssiutU, Assiut University
Other Study IDs: PEM in breast cancer
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PEM — Accuracy of PEM in detection of breast cancer

SUMMARY:
Investigate the accuracy of PEM in detection of breast cancer.

DETAILED DESCRIPTION:
Investigate the accuracy of positron emission mammography as non invasive method for early detection of breast cancer especially small sized cancers.

ELIGIBILITY:
Inclusion Criteria:

* patients suspected with breast cancer.

Exclusion Criteria:

* patient with glucose level >200 mg/dl.
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients suspected with breast cancer or pathological proven to have breast cancer, patients underwent breast mammography or breast US and suspected to have breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of positron emission mammography in breast cancer | Base line
  Investigate PEM as non invasive method for early detection of breast cancer

IPD SHARING:
Plan to Share IPD: Undecided